CLINICAL TRIAL: NCT02258126
Title: The Effect of Exercise on Hepatic Fat in Overweight Children; the EFIGRO Study
Brief Title: Effect of Exercise on Hepatic Fat in Overweight Children
Acronym: EFIGRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, IDOIA LABAYEN, Lecturer of Nutrition and Food Sciences, University of the Basque Country (UPV/EHU)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI13/01335
Record Dates: First submitted 2014-10-03; First posted 2014-10-07 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Non-alcoholic Fatty Liver Disease; Obesity; Metabolic Syndrome
Keywords: overweight children; hepatic fat; exercise; nutritional education program; cardiometabolic risk
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): healthy lifestyle education including healthy lifestyle education, supportive therapy and behavioral advice for both children and parents to improve nutrition and physical activity
  Interventions: Other: Multidisciplinary intervention program
- Exercise group (Experimental): multidisciplinary intervention program including healthy lifestyle education, supportive therapy and behavioral advice for for both children and parents to improve nutrition and physical activity and supervised exercise.
  Interventions: Other: Multidisciplinary intervention program

INTERVENTIONS:
Other: Multidisciplinary intervention program — Exercise group:
  The intervention program includes an education program promoting healthy dietary habits and physical activity (nutritionist), supportive therapy and behavioral advice for the family to improve nutrition and physical activity (psychologist) (2 times/month, for children and parents) and supervised exercise (3 times/week, 90 mins) program for 6 months.

SUMMARY:
The objective of the present study is to evaluate the effect of 6 months exercise intervention program on hepatic fat fraction in overweight children.

Methodology: A total of 160 children, 9-11 years old, will be randomly assigned to control (N=80) or intervention (N=80) groups. Training sessions will include 90 minutes of exercise, comprising warm-up and skill development. The control group will attend a healthy lifestyle education program (2 days/month) and the intervention group an exercise (3 days/week) and healthy lifestyle education (2 days/month) combined program. Before and after the intervention (6 months) hepatic fat fraction, body composition, , and cardiometabolic risk factors will be measured. Furthermore, dietary habits and physical activity, blood pressure and pubertal development will be evaluated before and after the intervention.

DETAILED DESCRIPTION:
The control group will attend a healthy lifestyle education program (2 days/month) and supportive therapy and behavioral advice for both children and parents to improve nutrition and physical activity (nutritionists and psychologists).

The intervention group will attend an exercise (3 days/week) and healthy lifestyle education (2 days/month) combined program. Training sessions will include 90 minutes of exercise, comprising warm-up and skill development, moderate to vigorous aerobic activities, flexibility and strength exercises.

Before (baseline) and after the intervention (6 months) total and abdominal adiposity, lean tissue mass and bone mass density (dual-X-ray-absorptiometry), abdominal visceral and hepatic adiposity (magnetic resonance imaging), and blood insulin, glucose, C-reactive protein, alanine aminotransferase, aspartate aminotransferase, gamma-glutamil transpeptidase and lipid profile will be measured. Furthermore, cardiorespiratory fitness (treadmill test) and blood pressure will be measured before and after the intervention. Changes (6 months - baseline) in dietary habits will be estimated by using two repeated 24h recalls and food frequency questionnaires and changes (6 months - baseline) in physical activity by accelerometry.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity status
* 9-11 years old

Exclusion Criteria:

* Medical conditions that hamper their participation in the exercise program
* Secondary obesity

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
changes in hepatic fat | baseline and 6 months
  Changes in hepatic fat fraction measured by magnetic resonance imaging after the 6 months intervention program

SECONDARY OUTCOMES:
Changes in Insulin sensitivity | baseline and 6 months
  Changes in insulin sensitivu¡ity measured by homeostasis model assessment (HOMA) after the 6 months intervention program
Changes in serum lipid profile | baseline and 6 months
  Changes in total, LDL- and HDL-cholesterol after the 6 months intervention program
Changes in liver enzymes | baseline and 6 months
  Changes in total, alanine transaminase (ALT), aspartate transaminase (AST) and gamma-GT after the 6 months intervention program
Changes in dietary habits | baseline and 6 months
  Changes in dietary habits estimated by 24h recall and food frequency questionnaire after the 6 months intervention program
Changes in physical activity | baseline and 6 months
  Changes in physical activity estimated by accelerometry after the 6 months intervention program
Changes in body composition | baseline and 6 months
  Changes in visceral adipose tissue (MRI), abdominal and total adiposity (DEXA), lean tissue mass and bone mass (DEXA) the 6 months intervention program
Changes in other cardiometabolic risk factors | baseline and 6 months
  Changes in blood pressure, leptin, adiponectin, C-reactive protein (CRP) after the 6 months intervention program

CONTACTS AND LOCATIONS:
Overall Officials: IDOIA LABAYEN, PhD, Principal Investigator — Department of Nutrition and Food Sciences, Faculty of Pharmacy, University of the Basque Country
Locations (1):
- Pediatric Endocrinology Unit of the University Hospital of Araba (HUA), Vitoria-Gasteiz, Araba, Spain

REFERENCES:
- [Background] Nobili V, Manco M. Therapeutic strategies for pediatric non-alcoholic fatty liver disease: a challenge for health care providers. World J Gastroenterol. 2007 May 14;13(18):2639-41. doi: 10.3748/wjg.v13.i18.2639. PMID 17552019
- [Result] Volovelsky O, Weiss R. Fatty liver disease in obese children--relation to other metabolic risk factors. Int J Pediatr Obes. 2011 Sep;6 Suppl 1:59-64. doi: 10.3109/17477166.2011.583661. PMID 21905818
- [Result] Welsh JA, Karpen S, Vos MB. Increasing prevalence of nonalcoholic fatty liver disease among United States adolescents, 1988-1994 to 2007-2010. J Pediatr. 2013 Mar;162(3):496-500.e1. doi: 10.1016/j.jpeds.2012.08.043. Epub 2012 Oct 17. PMID 23084707
- [Result] Kotronen A, Yki-Jarvinen H. Fatty liver: a novel component of the metabolic syndrome. Arterioscler Thromb Vasc Biol. 2008 Jan;28(1):27-38. doi: 10.1161/ATVBAHA.107.147538. Epub 2007 Aug 9. PMID 17690317
- [Result] Schwimmer JB, Pardee PE, Lavine JE, Blumkin AK, Cook S. Cardiovascular risk factors and the metabolic syndrome in pediatric nonalcoholic fatty liver disease. Circulation. 2008 Jul 15;118(3):277-83. doi: 10.1161/CIRCULATIONAHA.107.739920. Epub 2008 Jun 30. PMID 18591439
- [Result] Wicklow BA, Wittmeier KD, MacIntosh AC, Sellers EA, Ryner L, Serrai H, Dean HJ, McGavock JM. Metabolic consequences of hepatic steatosis in overweight and obese adolescents. Diabetes Care. 2012 Apr;35(4):905-10. doi: 10.2337/dc11-1754. Epub 2012 Feb 22. PMID 22357180
- [Result] Akin L, Kurtoglu S, Yikilmaz A, Kendirci M, Elmali F, Mazicioglu M. Fatty liver is a good indicator of subclinical atherosclerosis risk in obese children and adolescents regardless of liver enzyme elevation. Acta Paediatr. 2013 Mar;102(3):e107-13. doi: 10.1111/apa.12099. Epub 2012 Dec 29. PMID 23190373
- [Result] Davis CL, Pollock NK, Waller JL, Allison JD, Dennis BA, Bassali R, Melendez A, Boyle CA, Gower BA. Exercise dose and diabetes risk in overweight and obese children: a randomized controlled trial. JAMA. 2012 Sep 19;308(11):1103-12. doi: 10.1001/2012.jama.10762. PMID 22990269
- [Result] Escalante Y, Saavedra JM, Garcia-Hermoso A, Dominguez AM. Improvement of the lipid profile with exercise in obese children: a systematic review. Prev Med. 2012 May;54(5):293-301. doi: 10.1016/j.ypmed.2012.02.006. Epub 2012 Feb 23. PMID 22387009
- [Result] Koot BG, van der Baan-Slootweg OH, Tamminga-Smeulders CL, Rijcken TH, Korevaar JC, van Aalderen WM, Jansen PL, Benninga MA. Lifestyle intervention for non-alcoholic fatty liver disease: prospective cohort study of its efficacy and factors related to improvement. Arch Dis Child. 2011 Jul;96(7):669-74. doi: 10.1136/adc.2010.199760. Epub 2011 Apr 25. PMID 21518734
- [Result] Hallsworth K, Fattakhova G, Hollingsworth KG, Thoma C, Moore S, Taylor R, Day CP, Trenell MI. Resistance exercise reduces liver fat and its mediators in non-alcoholic fatty liver disease independent of weight loss. Gut. 2011 Sep;60(9):1278-83. doi: 10.1136/gut.2011.242073. Epub 2011 Jun 27. PMID 21708823
- [Result] Lee S, Bacha F, Hannon T, Kuk JL, Boesch C, Arslanian S. Effects of aerobic versus resistance exercise without caloric restriction on abdominal fat, intrahepatic lipid, and insulin sensitivity in obese adolescent boys: a randomized, controlled trial. Diabetes. 2012 Nov;61(11):2787-95. doi: 10.2337/db12-0214. Epub 2012 Jun 29. PMID 22751691
- [Result] Oh S, Tanaka K, Warabi E, Shoda J. Exercise reduces inflammation and oxidative stress in obesity-related liver diseases. Med Sci Sports Exerc. 2013 Dec;45(12):2214-22. doi: 10.1249/MSS.0b013e31829afc33. PMID 23698242
- [Derived] Labayen I, Cadenas-Sanchez C, Idoate F, Medrano M, Tobalina I, Villanueva A, Rodriguez-Vigil B, Alvarez de Eulate N, Oses M, Cabeza R. Liver Fat, Bone Marrow Adipose Tissue, and Bone Mineral Density in Children With Overweight. J Clin Endocrinol Metab. 2023 Dec 21;109(1):e253-e258. doi: 10.1210/clinem/dgad429. PMID 37490040
- [Derived] Cadenas-Sanchez C, Cabeza R, Idoate F, Oses M, Medrano M, Villanueva A, Arenaza L, Sanz A, Ortega FB, Ruiz JR, Labayen I. Effects of a Family-Based Lifestyle Intervention Plus Supervised Exercise Training on Abdominal Fat Depots in Children With Overweight or Obesity: A Secondary Analysis of a Nonrandomized Clinical Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2243864. doi: 10.1001/jamanetworkopen.2022.43864. PMID 36441551
- [Derived] Cadenas-Sanchez C, Idoate F, Cabeza R, Villanueva A, Rodriguez-Vigil B, Medrano M, Oses M, Ortega FB, Ruiz JR, Labayen I. Effect of a Multicomponent Intervention on Hepatic Steatosis Is Partially Mediated by the Reduction of Intermuscular Abdominal Adipose Tissue in Children With Overweight or Obesity: The EFIGRO Project. Diabetes Care. 2022 Sep 1;45(9):1953-1960. doi: 10.2337/dc21-2440. PMID 36044664
- [Derived] Medrano M, Arenaza L, Migueles JH, Rodriguez-Vigil B, Ruiz JR, Labayen I. Associations of physical activity and fitness with hepatic steatosis, liver enzymes, and insulin resistance in children with overweight/obesity. Pediatr Diabetes. 2020 Jun;21(4):565-574. doi: 10.1111/pedi.13011. Epub 2020 Apr 12. PMID 32237015
- [Derived] Medrano M, Arenaza L, Ramirez-Velez R, Ortega FB, Ruiz JR, Labayen I. Prevalence of responders for hepatic fat, adiposity and liver enzyme levels in response to a lifestyle intervention in children with overweight/obesity: EFIGRO randomized controlled trial. Pediatr Diabetes. 2020 Mar;21(2):215-223. doi: 10.1111/pedi.12949. Epub 2019 Dec 10. PMID 31778277
- [Derived] Labayen I, Medrano M, Arenaza L, Maiz E, Oses M, Martinez-Vizcaino V, Ruiz JR, Ortega FB. Effects of Exercise in Addition to a Family-Based Lifestyle Intervention Program on Hepatic Fat in Children With Overweight. Diabetes Care. 2020 Feb;43(2):306-313. doi: 10.2337/dc19-0351. Epub 2019 Jun 21. PMID 31227585
- [Derived] Medrano M, Cadenas-Sanchez C, Alvarez-Bueno C, Cavero-Redondo I, Ruiz JR, Ortega FB, Labayen I. Evidence-Based Exercise Recommendations to Reduce Hepatic Fat Content in Youth- a Systematic Review and Meta-Analysis. Prog Cardiovasc Dis. 2018 Jul-Aug;61(2):222-231. doi: 10.1016/j.pcad.2018.01.013. Epub 2018 Feb 13. PMID 29452135
- [Derived] Nystrom CD, Henriksson P, Martinez-Vizcaino V, Medrano M, Cadenas-Sanchez C, Arias-Palencia NM, Lof M, Ruiz JR, Labayen I, Sanchez-Lopez M, Ortega FB. Does Cardiorespiratory Fitness Attenuate the Adverse Effects of Severe/Morbid Obesity on Cardiometabolic Risk and Insulin Resistance in Children? A Pooled Analysis. Diabetes Care. 2017 Nov;40(11):1580-1587. doi: 10.2337/dc17-1334. Epub 2017 Sep 22. PMID 28939688